CLINICAL TRIAL: NCT05695872
Title: The Best Approach to Zygomaticomaxillary Fractures: A Comparison of Three Surgical Approaches
Brief Title: A Comparison of Three Surgical Approaches to Zygomaticomaxillary Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Lydia Nabil, Associate Professor of Oral and Maxillofacial Surgery, University of Alexandria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UAlexandriaMaxFacSurg
Record Dates: First submitted 2023-01-11; First posted 2023-01-25 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Zygomatic Fractures
MeSH Terms: conditions — Zygomatic Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- subtarsal approach (Active Comparator)
  Interventions: Procedure: subtarsal approach
- conventional transconjunctival approach (Active Comparator)
  Interventions: Procedure: conventional transconjunctival approach
- transconjunctival approach with Y- modification (Active Comparator)
  Interventions: Procedure: transconjunctival approach with Y- modification

INTERVENTIONS:
Procedure: subtarsal approach — surgical approach
  Arms: subtarsal approach
Procedure: conventional transconjunctival approach — surgical approach
  Arms: conventional transconjunctival approach
Procedure: transconjunctival approach with Y- modification — surgical approach
  Arms: transconjunctival approach with Y- modification

SUMMARY:
The study is a randomized controlled clinical trial, following the Consolidated Standards of Reporting Trials (CONSORT) guidelines. The study is intended to compare between the subtarsal approach, conventional transconjuctival approach and the Y- modification of the transconjuctival approach in the management of zygomatico-maxillay complex fracture.

DETAILED DESCRIPTION:
The study is a randomized controlled clinical trial. Twenty-four patients with age range of 20-50 years requiring open reduction and fixation of a fractured zygomatic complex were randomly divided into three equal groups according to the approach used:

Group A: subtarsal approach group. Group B: conventional transconjuctival approach group. Group C: Y- modification of the transconjuctival approach group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ZMC fractures requiring open reduction and internal fixation.
* Adult patients aged between 20 and 50 years with no gender predilection.

Exclusion Criteria:

* An existing laceration in the inferior and lateral periorbital site.
* Infection at the fracture line.
* Comminuted fracture with bone loss.
* Acute and chronic conjunctival diseases.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-08-26 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-05 (Actual)

PRIMARY OUTCOMES:
accessibility to the fracture site | intraoperative
  Adequate exposure provided by the incision and accessiblity to proper fracture reduction and fixation was assigned as Yes or No
esthetic appearance and scarring | 6 weeks postoperative
  Postoperative scarring was recorded as noticeable or unnoticeable
radiographic verification of adequacy of fracture reduction | immediate postoperative
  computed tomography was requested for adequacy of fracture reduction assessment and this outcome was assigned as Yes or No

SECONDARY OUTCOMES:
The duration for exposure of the fracture site | intraoperative
  The duration from performing the incision till the field exposure calculated in minutes
postoperative pain | at 24 hours and 1 week
  Pain was evaluated at 24 hours and at 1 week according to a 10-point Visual Analogue Scale (VAS), (0-1=none,2-4=mild,5-7=moderate,8-10=severe).
sensory nerve function | 3 months postoperative
  Subjective assessment of the infraorbital nerve sensation by patient questioning about any alteration in sensation at 3 months postoperatively.
  Objective assessment by dental probe pressure to assess sensory changes along the distribution of the infraorbital nerve with contralateral side comparison

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Melek LN, Noureldin MG. Zygomaticomaxillary complex fractures: finding the least complicated surgical approach (A Randomized Clinical Trial). BMC Oral Health. 2023 Aug 4;23(1):539. doi: 10.1186/s12903-023-03249-8. PMID 37542217